CLINICAL TRIAL: NCT01020708
Title: A Phase I Double-blind, Randomized, Comparator-controlled Study of the Safety and Tolerability of N-acetylcysteine Plus Mesalamine Enema in Subjects With Left-sided Ulcerative Colitis
Brief Title: Study of the Safety and Tolerability of ALTH12 Versus Mesalamine Enema in Subjects With Left-Sided Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altheus Therapeutics, Inc. (Industry)
Responsible Party: Richard F. Harty, M.D., Altheus Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALTH12-003
Record Dates: First submitted 2009-11-20; First posted 2009-11-24 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Ulcerative Colitis
Keywords: colitis; inflammatory bowel disease; ulcerative colitis; rectal administration; enema; mesalamine
MeSH Terms: conditions — Colitis, Ulcerative; Colitis; Inflammatory Bowel Diseases | interventions — Mesalamine; Acetylcysteine; Enema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Comparator (Active Comparator): Mesalamine enema
  Interventions: Drug: mesalamine
- ALTH12-1:4 (Experimental): ALTH12-1:4 experimental treatment dose
  Interventions: Drug: ALTH12-1:4
- ALTH12-2:4 (Experimental): ALTH12-2:4 experimental treatment dose
  Interventions: Drug: ALTH12-2:4

INTERVENTIONS:
Drug: mesalamine — 4.0g mesalamine rectal suspension, rectally administered enema, 60ml volume, 4.0g mesalamine, once daily
  Other Names: Rowasa; 5-ASA; 5-aminosalicylic acid
  Arms: Comparator
Drug: ALTH12-1:4 — ALTH12-1:4 rectal suspension, rectally administered enema, 60mL volume, 4.0g mesalamine, 1.0g N-acetylcysteine
  Other Names: mesalamine; 5-ASA; N-acetylcysteine; NAC; enema
  Arms: ALTH12-1:4
Drug: ALTH12-2:4 — ALTH12-2:4 rectal suspension, rectally administered enema, 60mL volume, 4.0g mesalamine, 2.0g N-acetylcysteine
  Other Names: mesalamine; 5-ASA; N-acetylcysteine; NAC
  Arms: ALTH12-2:4

SUMMARY:
This Phase I study will be a closely monitored trial of a small number of subjects to establish, preliminarily, the tolerability and safety of two ALTH12 enema formulations: ALTH12-1:4 and ALTH12-2:4. The study will be conducted in two parts. The first part will be the assessment of the safety and tolerability of a single dose of ALTH12-1:4 or the comparator, mesalamine (4.0g 5-ASA) followed by an assessment of repeated administrations of study drug (ALTH12-1:4 or comparator) for 6 weeks. The second part will be the same assessment for ALTH12-2:4. Three subjects will be enrolled in each cohort: 2 to receive ALTH12 enema therapy and 1 subject to receive comparator enema therapy. A total of up to 9 patients will be enrolled in this study, allowing for up to 3 replacement or additional patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects are eligible if they are ≥ 18 years of age and ≤ 64 years
* They have a documented history of idiopathic ulcerative colitis based on endoscopic and/or histologic findings involving the left side of the colon, with mild active disease or disease in remission.
* Eligible subjects will have a documented history of ulcerative colitis, and a modified UCDAI with a sigmoidoscopy score of 1 point or less and Physician's rating of disease score of 1 point or less (mild or remission).
* Laboratory data:

  1. White blood cell count between 4,500 and 10,000 cells/mL
  2. Platelet count: 150,000-450,000 cells/mL
  3. Hemoglobin > 10.0 g/dL
  4. Total bilirubin < 1.5 mg/dL
  5. Aspartate aminotransferase < 100 u/dL
  6. Alanine aminotransferase < 100 u/dL
  7. Alkaline phosphatase < 250 u/dL
  8. Blood urine nitrogen < 40 mg/dL
  9. Creatinine < 1.5 mg/dL
  10. Amylase < 150 U/L
* Satisfied one of the following:
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening; surgically sterile, post-menopausal, abstinent, or patient or partner agree to use a medically appropriate form of birth control from screening to until 1 month after the last dose of study medication.
* Male subjects must be surgically sterile, abstinent, or patient or partner compliant with a contraceptive regimen from screening to until 1 month after the last dose of study medication.
* They are able to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.

Exclusion Criteria:

Subjects will be excluded if:

* They have documented history of proctitis or active proctitis confined to 15cm or less from the anal verge.
* They demonstrate signs and symptoms of fulminant colitis, bowel stricture, toxic megacolon, an anticipated need for blood transfusion for gastrointestinal bleeding, or demonstrate evidence of peritonitis.
* They receive a Physician's rating of disease severity as part of the modified UCDAI of 2 or greater (moderate or severe disease) or an endoscopy score of 2 or greater.
* They have shown evidence of high grade dysplasia on endoscopic examinations.
* Their stool contains enteric pathogens or Clostridium difficile toxins.
* They have a history of recurrent Clostridium difficile infection.
* They have prior history of biologic therapy.
* They have received systemic steroids or immunosuppressants within the previous 4 weeks.
* Treatment in the last 2 weeks that included antibiotic, antifungal, antiparasitic medications, or rectally administered steroids (e.g. Cortenema®) and/or 5-ASA enema (e.g. Rowasa®).
* They have a history of cancer (defined as malignancy within 5 years except for squamous cell or basal cell cancers of the skin), asthma, or bronchospasm.
* Positive pregnancy test or lactating subjects.
* There is evidence of chemical abuse.
* They have a known allergy to N-acetylcysteine or Mesalamine.
* They have a history of failure to retain enemas.
* Other clinically significant diseases that could interfere with the protocol compliance appear. These would include clinically important hematological, renal, hepatic, metabolic, psychiatric, central nervous system (CNS), pulmonary or cardiovascular disease.
* Any condition which the study physician judges to preclude safe participation in the study or to confound the evaluation of the study outcome.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of ALTH12 when given by intrarectal administration over 6 weeks to subjects with ulcerative colitis (UC) involving the left side of the colon | 6 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philip B Miner, M.D., Principal Investigator — Oklahoma Foundation for Digestive Research
Locations (1):
- Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma, United States